CLINICAL TRIAL: NCT02122484
Title: Study of Anti-inflammatory Treatment With Colchicine in Patients Undergoing Elective Coronary Artery Bypass Graft Surgery to Reduce Reperfusion Damage
Brief Title: Colchicine in Coronary Artery Bypass Graft (CABG)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: G.Gennimatas General Hospital (Other)
Collaborators: Evangelismos Hospital (Other)
Responsible Party: Principal Investigator, Spyridon Deftereos, Director, Cardiac Catheterization Department, G.Gennimatas General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COL.CABG
Record Dates: First submitted 2014-04-22; First posted 2014-04-24 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Elective Coronary Artery Bypass Graft Surgery
Keywords: reperfusion damage
MeSH Terms: conditions — Reperfusion Injury | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Placebo Comparator): Patients taking placebo
- Colchicine (Experimental): Active treatment group
  Interventions: Drug: Colchicine

INTERVENTIONS:
Drug: Colchicine — colchicine p.os 0.5 mg bid for two days before undergoing elective CABG surgery and eight days after the operation
  Arms: Colchicine

SUMMARY:
There is evidence that inflammatory processes may play a key role during surgical myocardial reperfusion. The hypothesis of this study is that colchicine, an anti-inflammatory agent, may lead to reduction in periprocedural infarct size, when administered during elective coronary artery bypass graft surgery.

ELIGIBILITY:
Inclusion Criteria:

* The study will enroll patients 18 years old or older who are eligible to undergo CABG surgery.

Exclusion Criteria:

Excluded are patients:

* with age > 80 years old
* scheduled for concomitant valve surgery
* scheduled for coronary surgery without cardiopulmonary bypass
* with peripheral vascular disease aﬀecting the upper limbs
* with acute coronary syndrome within the previous 4 weeks
* on inotropic or mechanical circulatory support before induction of anaesthesia
* with any disorder that could potentially increase preoperative cTnI concentrations (eg, percutaneous coronary intervention within the previous 6 weeks)
* with active inflammatory diseases, infectious diseases or known malignancy
* under treatment with corticosteroids, anti-inflammatory agents or disease modifying agents
* with known hypersensitivity-allergy to colchicine
* under chronic treatment with colchicine
* with severe renal failure (eGFR < 35 ml/min/1.73 m2)
* with hepatic failure (Child - Pugh class B or C)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-11; Primary Completion 2014-06 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Myocardial damage marker levels | Days 1-2 post-CABG

SECONDARY OUTCOMES:
All cause mortality | At one and at six months after CABG

CONTACTS AND LOCATIONS:
Overall Officials: Spyridon Deftereos, MD, Principal Investigator — Athens General Hospital "G. Gennimatas"
Locations (1):
- Athens General Hospital "G. Gennimatas", Athens, Attica, Greece

REFERENCES:
- [Derived] Giannopoulos G, Angelidis C, Kouritas VK, Dedeilias P, Filippatos G, Cleman MW, Panagopoulou V, Siasos G, Tousoulis D, Lekakis J, Deftereos S. Usefulness of colchicine to reduce perioperative myocardial damage in patients who underwent on-pump coronary artery bypass grafting. Am J Cardiol. 2015 May 15;115(10):1376-81. doi: 10.1016/j.amjcard.2015.02.036. Epub 2015 Feb 18. PMID 25784519